CLINICAL TRIAL: NCT06075680
Title: Effect of Non-Surgical Periodontal Treatment on Inflammasome-Related Proteins in Periodontal Diseases
Brief Title: Effect of Periodontal Treatment on Inflammasome Proteins in Periodontal Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDK-2022-10763
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Periodontal Diseases; Gingivitis; Periodontitis
Keywords: Periodontitis; Inflammasomes; Gingivitis
MeSH Terms: conditions — Periodontal Diseases; Gingivitis; Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy (No Intervention): Periodontally healthy patients received no intervention.
- Gingivitis (Active Comparator): Gingivitis group received Non-Surgical Periodontal Treatment. They received Scaling and Root Planning procedure with ultrasonic scalers and hand curettes. The entire non-surgical periodontal treatment of gingivitis groups was completed in a total of 2 sessions in a week.
  Interventions: Procedure: Non-Surgical Periodontal Treatment
- Stage III Grade C Periodontitis (Active Comparator): Stage III Grade C group received Non-Surgical Periodontal Treatment. They received Scaling and Root Planning procedure with ultrasonic scalers and hand curettes. The patients were subjected to quadrant-wise full-mouth subgingival scaling and root planning under local anesthesia. The entire non-surgical periodontal treatment of periodontitis groups was completed in a total of 4 sessions in two weeks.
  Interventions: Procedure: Non-Surgical Periodontal Treatment

INTERVENTIONS:
Procedure: Non-Surgical Periodontal Treatment — The primary goal of nonsurgical periodontal therapy is to control microbial periodontal infection by removing bacterial biofilm, calculus, and toxins from periodontally involved root surfaces. Performing a thorough periodontal debridement under local anesthesia will stop disease progression and result in improvement in the clinical signs and symptoms of active disease
  Arms: Gingivitis; Stage III Grade C Periodontitis

SUMMARY:
The present study aimed to assess the effect of non-surgical periodontal treatment on serum and salivary IL-1beta, IL-18, NLRP3, ASC and Caspase-1 levels in gingivitis and Stage III Grade C periodontitis. 15 periodontally healthy, 15 gingivitis and 15 Stage III Grade C periodontitis patients were enrolled. At baseline, serum and saliva samples were collected and the whole mouth clinical periodontal parameters were recorded. Periodontitis and gingivitis patients received non-surgical periodontal treatment. Clinical parameters were re-measured and samples were re-collected at 1 and 3 months after treatment. Serum and salivary protein levels were analyzed by ELISA. Data were analyzed using appropriate statistical tests.

DETAILED DESCRIPTION:
New insights into the first line of immune response to infection and stress signals at the cellular level have reported the participation of cytoplasmic nucleotide-binding domain-like receptors containing multi-protein complexes named inflammasomes. The inflammasomes play a key role in innate immunity by regulating maturation of proinflammatory cytokines of the interleukin 1beta and 18. The inflammasome depends on assembly of a sensor, for instance nod-like receptor family pyrin domaincontaining protein (NLRP), with an adaptor,apoptosis-associated speck-like protein containing a caspase recruitment domain (ASC), allowing recruitment and activation of an inflammatory caspase-1. Although different inflammasomes have been described, the NLRP3/ASC/caspase-1 multi-protein complex, known as NLRP3 inflammasome, has been most intensively studied.

Sample size was calculated based on a previous study concerning levels of inflammasome complex proteins in periodontal diseases.To maintain estimates at an optimal level of precision,minimize impact of exclusions and dropouts, and establish significant differences in results at a 95% confidence level, alfa value=0.05, and 83% power.Therefore, the study sample included a total of 45 patients( 15 periodontally healthy, 15 gingivitis, 15 sStage III Grade C Periodontitis). The whole mouth clinical periodontal examination included measurement of probing depth (PPD), clinical attachment level (CAL), presence of bleeding on probing (BOP), gingival index (GI), and plaque index (PI) at 6 sites per tooth, except the third molars. The presence and type of the alveolar bone loss were assessed on the digital panoramic radiograph in each participant, which was supplemented with periapical radiographs if necessary. Periodontal status of each patient was evaluated by a single calibrated periodontists with a manual probe. The diagnosis of periodontitis or periodontally health was determined according to the 2017 World Workshop on Classification of Periodontal and Peri-Implant Diseases and Conditions. Periodontally healthy individuals (n=15) in the control group had no sites with PD >3 mm and CAL >2 mm and also no radiographic evidence of alveolar bone loss. BOP was <10% in the whole mouth. Healthy group also exhibited no history of periodontitis. Gingivitis patients had PD≤3 mm, intact periodontium, no destruction in alveolar bone radiographically and BOP>10%. Stage III grade C patient had clinical attachment loss (CAL)≥ 5, radiographic bone loss (RBL) extending to the middle third of root and beyond, ≤ 4 tooth loss due to periodontitis, percentage of bone loss by age is >1.

Treatment The recruited periodontitis and gingivitis patients received conventional quadrant scaling and root planning (SRP). SRP was performed by the same clinician using ultrasonic inserts and manual periodontal curettes. Re-evaluations were performed at 1 and 3 months following the completion of the SRP. No periodontal intervention was carried out in the periodontally healthy controls.

Saliva and Serum Sampling A total of 5 mL of unstimulated whole saliva was collected by passive drool method between 9:00 and 10:00 am. The participants were advised to avoid food consumption for three hours before sample collection. The participants were seated upright and saliva was collected over a period of 5 minutes with instructions to pool saliva in the floor of the mouth and passively drool it into a sterile glass beaker. The saliva samples were centrifuged at 5000 rpm for 10 minutes at room temperature, and supernatants were collected and stored at -80°C. A total of 5 mL of blood was collected from the antecubital fossa by venepuncture method. Serum was isolated from the blood by centrifuging at 3000 rpm for 20 minutes followed by its rapid transfer to a sterile polypropylene tube and storage at -80°C.

Biomarker Immunoassays: Serum and salivary samples of IL-1beta, IL-18, NLRP3, ASC and Caspase-1 were measured by ELISA using commercial kits.

Statistical Analysis All statistical analyses were carried out with the standard statistical software package. For the intra-group comparisons, if the data were not normally disturbed, Friedman test and the Dunn test with the Bonferroni correction were used to analyze the change between baseline and 1 month and 3 months after treatment. For inter-group comparisons, Mann-Whitney U test for normally and non-normally disturbed data. The Spearman's rank correlation test was used to detect the correlations of biochemical parameters with clinical parameters and each others in diseased group before and after treatment. All tests were performed at significance level of P <0.05.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy and non-smoker individuals
* having ≥20 teeth present (except third molars)
* individuals with periodontally healthy, gingivitis or stage III grade C periodontitis diagnoses

Exclusion Criteria:

* having any diagnosed medical disorders such as diabetes mellitus, cardiovascular diseases, rheumatoid arthritis...
* usage of antibiotics, non-steroidal anti-inflammatory drugs and immunosuppressive agents within the past 6 months.
* periodontal treatment within the preceding 6 months.
* pregnant/ lactating/ postmenopausal females.
* Current orthodontic treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Salivary NLRP3 levels (ng/ml) | from baseline to 1 month and 3 months after treatment
  change in salivary NLRP3 levels from baseline to 1 month and 3 months after treatment
Salivary ASC levels (pg/ml) | from baseline to 1 month and 3 months after treatment
  change in salivary ASC levels from baseline to 1 month and 3 months after treatment
Salivary Caspase-1 levels (ng/ml) | from baseline to 1 month and 3 months after treatment
  change in salivary Caspase-1 levels from baseline to 1 month and 3 months after treatment
Salivary IL-1beta levels (pg/ml) | from baseline to 1 month and 3 months after treatment
  change in salivary IL-1beta levels from baseline to 1 month and 3 months after treatment
Salivary IL-18 levels (pg/ml) | from baseline to 1 month and 3 months after treatment
  change in salivary IL-18 levels from baseline to 1 month and 3 months after treatment

SECONDARY OUTCOMES:
Serum NLRP3 levels (ng/ml) | from baseline to 1 month and 3 months after treatment
  change in serum NLRP3 levels from baseline to 1 month and 3 months after treatment
Serum ASC levels (pg/ml) | from baseline to 1 month and 3 months after treatment
  change in serum ASC levels from baseline to 1 month and 3 months after treatment
Serum Caspase-1 levels (ng/ml) | from baseline to 1 month and 3 months after treatment
  change in serum Caspase-1 levels from baseline to 1 month and 3 months after treatment
Serum IL-1beta levels (pg/ml) | from baseline to 1 month and 3 months after treatment
  change in serum IL-1beta levels from baseline to 1 month and 3 months after treatment
Serum IL-18 levels (pg/ml) | from baseline to 1 month and 3 months after treatment
  change in serum IL-18 levels from baseline to 1 month and 3 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No